CLINICAL TRIAL: NCT06651164
Title: Psychosomatic Risk Screening in the Inpatient Care of Physically Ill Patients: a Feasibility Study
Brief Title: Psychosomatic Risk Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hans-Christoph Friederich, Prof. Dr. Hans-Christoph Friederich, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: S-301/2024
Record Dates: First submitted 2024-07-22; First posted 2024-10-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
Keywords: psychosocial risk factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: psychosocial risk screening conducted (Experimental): Patients in the intervention group are interviewed during admission on possible risk factors using the tablet-based screening questionnaire. The survey takes about 10 minutes. Once the screening has been completed, the results are immediately evaluated electronically and can be viewed by the person carrying out the screening. The patient is informed of the result (conspicuous/not conspicuous). If the psychosomatic screening is positive, the patient is asked if she/he is willing to be visited by a psychosomatic consultant. This contact will last about 15-45 minutes. If the social services screening is positive, the social services will introduce themselves in any case. Depending on the needs for regulation or counseling, this will result in a contact of 10-45 minutes. We use established and validated metrics and questionnaires.
  Interventions: Diagnostic Test: psychosocial risk screening
- Control: psychosocial risk screening is not conducted (No Intervention): Patients assigned to the control group will be treated as usual. Besides medical treatment this may also include consultations from a psychosomatic specialist and/or a social worker if the patient asks for it or the staff deems it necessary.

INTERVENTIONS:
Diagnostic Test: psychosocial risk screening — * combined tablet-based screening questionnaire for psychosomatic screening and social service screening
  * in case of positive psychosomatic or social service screening subsequent psychosomatic and / or social service consultation
  Arms: Intervention: psychosocial risk screening conducted

SUMMARY:
Mental health problems are common in terms of lifetime prevalence and often occur in combination with chronic physical illnesses. It is therefore reasonable to assume that there is considerable mental health comorbidity among inpatients. A recent retrospective analysis of patient data from a tertiary care internal medicine clinic also showed that the length of stay in hospital was longer for patients with mental comorbidity. This effect was particularly pronounced in the case of severe physical multimorbidity.

Our hypothesis is that the implementation of psychosocial risk screening as part of the inpatient admission process is suitable to identify the need for psychosomatic and social service counselling and treatment at an early stage and to address it appropriately from a medical, psychological and social service perspective in order to reduce the length of inhouse treatment.

Two consecutive studies are planned to test this hypothesis. The present study is a randomised feasibility study. Patients will be enrolled and assigned to the intervention or control group. Only the intervention group will receive screening. The psychosomatic and social screening will be differentiated according to previously defined risk categories. In some cases, established standardised questionnaires (PHQ-4, Audit-C, Clinical Frailty Scale, Six Item Screener) are used. In other cases, we have developed our own questions. Patients are screened by physicians or students in their practical year when they are admitted to our pilot ward. If the psychosomatic screening is positive and the patient agrees, they are referred to the psychosomatic consultation service. If the social service screening is positive, the patient will be seen by the social service.

The main objective of this study is to obtain informed consent from 30% of the eligible patients as a parameter for the feasibility and acceptance of such screening within an integrated psychosomatic and social service care concept. A study period of 3 months is planned for the feasibility study. The feasibility study will be analysed using descriptive statistics. The main study, which has not yet been applied for, is planned as a randomised intervention study. The main objective criterion will be to reduce the length of stay through screening and, if necessary, timely psychosomatic or social counselling.

DETAILED DESCRIPTION:
Mental health problems are common in terms of lifetime prevalence and often occur in combination with chronic physical illnesses. Mental comorbidities in physically ill patients lead to higher morbidity and mortality, greater demands on the healthcare system and higher treatment costs.

Among medical inpatients it can therefore be assumed that there is considerable mental comorbidity. In a large retrospective analysis of around 28,500 patient data sets from the Department of Internal Medicine at Heidelberg University Hospital, we could show that the length of stay in hospital for patients with mental comorbidity was extended by a total of 2 days when compared with patients who had no documented mental comorbidity. This effect was particularly pronounced in the case of major physical multimorbidity. In addition to previously documented psychiatric and psychosomatic diseases, there is a tremendous lack of recognition and diagnosis of relevant mental comorbidities. It has also been shown that other non-acute medical factors, such as functional limitations, impairment of activities of daily living, frailty, cognitive limitations or the lack of a receiving care facility, prolong the length of stay.

To address these problems in health care, some guidelines recommend systematic screening for mental and functional risk-factors, but still this has not been implemented in routine inpatient medical wards. The implementation of psychosomatic risk screening as part of the inpatient admission process could be suitable for detecting the need for psychosomatic and social service at an early stage and addressing it accordingly with psychotherapy, psychopharmacy and qualified social support. It may also be possible to reduce the length of stay in hospital. In this pilot project, a psychosocial risk screening with subsequent psychosomatic assessment by a consultant and introduction to social services is to be evaluated with regard to the feasibility of integration into ward procedures and acceptance by patients. The study is designed as a randomized feasibility study. Patients are included in the study on admission to a medical ward and randomly assigned to the intervention or the control group. The intervention group receives the screening and if necessary subsequent further care, the control group does not receive screening.

Screening focuses on previously defined psychosocial risk categories:

As part of the psychosomatic screening, the risk categories of sleep disorder and psychotropic drug use, depression, anxiety disorder, subjective disease burden, risky alcohol consumption, frailty and cognitive impairment are examined based on previous results.

For the social services screening, relevant consultation and intervention needs such as a general need for advice on social law issues, a lack of health insurance, a lack of financial security, the presence of a legal guardian, a need for care at home, an existing or possibly increased level of care and interest in follow-up treatment or rehabilitation measures are queried.

In the event of a conspicuous psychosomatic screening, a consecutive assessment is carried out by a psychosomatic consultant if consent is given. In the event of a conspicuous social services screening, a social worker is called. If the screening is negative, there will be no further assessment or consultation by the respective services at this time.

The current study serves to prepare a larger randomized trial to test the effect of a psychosocial risk screening together with a defined care path on the reduction of length of stay in patients with medical diseases.

ELIGIBILITY:
Inclusion Criteria:

* The target group are all adult (age >=18 years) physically ill patients capable of giving consent on the pilot ward.

Exclusion Criteria:

* Acute mental illnesses that require immediate further treatment (e.g., active suicidal ideation, acute psychotic state)
* The length of stay is too short to carry out a psychosomatic and/or a social services consultation. This can be assumed if the expected length of stay is less than or equal to three days.
* Insufficient knowledge of the German language.
* Cognitive impairment or significant hearing impairment that makes it impossible for the person carrying out the screening and answering the questions adequately.
* in case of re-admission if patient has already been included in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Acceptance of study participation | On admission day (day 1) or first possible day of patient consultation
  The main target criterion of the feasibility study is the rate of patients accepting study We will determine the rate of eligible patients accepting study participation as the main target criterion of the feasibility study.

SECONDARY OUTCOMES:
Compliance with screening procedure/ result | At day 1 /day of risk screening
  We will determine the rate of screening results that are implemented accordingly by the staff (psychosomatic consultation, social service consultation)
Compliance with screening recommendations | At day 1 /day of risk screening
  We will determine the rate of study patients willing to meet with a psychosomatic consultant and / or social worker, if indicated by risk screening
Loss to follow up | 3 month after discharge from the ward
  We will determine the rate of study participants with completed follow up assessment
Compliance with all study procedures | 3 month after discharge from the ward
  We will determine the rate of study patients with fully completed study procedures (electronic risk screening, consultation with psychosomatic expert and / or social worker, follow up assessment)
Patient's physical health at the time of follow up | 3 month after discharge from the ward
  We will determine physical health using a visual analogue scale (VAS)
Patient's general wellbeing at the time of follow up | 3 month after discharge from the ward
  We will determine general wellbeing using a visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Friederich, Prof. Dr., Principal Investigator — Heidelberg University Clinic - Department for general internal medicine and psychosomatics
Locations (1):
- Heidelberg University Clinic - Medical Clinic, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stahl-Toyota S, Nikendei C, Nagy E, Bonsel S, Rollmann I, Unger I, Szendrodi J, Frey N, Michl P, Muller-Tidow C, Jager D, Friederich HC, Hochlehnert A. Interaction of mental comorbidity and physical multimorbidity predicts length-of-stay in medical inpatients. PLoS One. 2023 Jun 22;18(6):e0287234. doi: 10.1371/journal.pone.0287234. eCollection 2023. PMID 37347745